CLINICAL TRIAL: NCT04989582
Title: Effectiveness of a Nursing Intervention for Nurses Have Experienced Trauma: a Study Based on Swanson's Caring Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Y-2019-0083
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Nurses Who Have Experienced Trauma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing intervention (Experimental): Nurses randomly assigned by applying a random selection method
  Interventions: Other: The trauma recovery nursing intervention program
- No intervention (No Intervention): Nurses randomly assigned by applying a random selection method

INTERVENTIONS:
Other: The trauma recovery nursing intervention program — The trauma recovery nursing intervention program was for adults who had experienced trauma and consisted of eight sessions, each lasting 30 min. It included a spoken audio track that was accompanied by visual prompts to provide knowledge on traumatic stress and introduce trauma recovery methods. Its online format made it convenient and widely accessible, and allowed for a low-intensity, cost-effective educational program. The program focused on providing self-help guidelines for clients to develop their mental and physical well-being.
  Arms: Nursing intervention

SUMMARY:
This study aimed to (1) develop an internet-based psychiatric nursing intervention, based on Swanson's theory of caring, and (2) examine its effects on functional health, resilience, social support, post-traumatic stress, depression, and anxiety.

This study was a randomized clinical trial(RCT) study with repeated measures to identify the effectiveness of an internet-based psychiatric nursing intervention. Participants were evaluated at the following time points: pre-test (pre), post-test (post-test 1, immediately after intervention), and follow-up (post-test 2, one month after the intervention) to assess the sustainability of the internet-based psychiatric nursing intervention.

Of the 112 women who enrolled in the study, 10 dropped out before post-test 1, resulting in 102 participants who completed all interventions and surveys.

ELIGIBILITY:
Inclusion Criteria:

1. nurse aged from 23 to 40 years
2. a PTS score of 64 or lower on the PTSD checklist for DSM-5 (PCL-5) developed by Weathers et al., revised by Weathers et al., and translated into Korean by Kim et al.,
3. nurse who can access the program through a computer or mobile
4. nurse who understand the purpose of the research and voluntarily agree to participate in the research.

Exclusion Criteria:

1. presence of psychiatric conditions with hallucinations and delusions
2. diagnosis of an intellectual disability that would make understanding the intervention procedure difficult. Although a standard cut-off was not present in the PCL-5, women who exceeded 80% (64 points) of the total score were excluded to rule out high-risk women with severe trauma.

Ages: 23 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
functional health | one month after the intervention
  The Functional Health Pattern Assessment Screening Tool (FHPAST) was developed by Jones (2002) and adapted by Keum and Kim (2012). The FHPAST is a self-report scale consisting of 58 items, each with a 4-point scale (1 to 4). Sixteen questions (43-58) are reverse scored. Mean scores of three or higher indicate that the physiological-spiritual function is at a healthy level and the individual is ready for health promotion. In the Jones study (2002), the reliability was Cronbach's α = .70 and .90.
resilience | one month after the intervention
  Resilience was assessed using the Korean version of the Resilience Scale (K-CD-RISC) developed by Connor and Davidson (2003) and standardized by Baek, Lee, Joo, Lee, and Choi (2010). This selfreported instrument consists of 25 items scored on a 5-point scale ranging from 0 (not at all) to 4 (almost always). The scale comprises five factors: hardiness, persistence, optimism, support, and spirituality. Scores range from 0 to 100, with higher scores indicating higher levels of resilience. The Cronbach's α was 0.89 in a previous study (Connor & Davidson, 2003).
social support | one month after the intervention
  Social support was measured using the Social Provisions Scale (SPS), developed by Cutrona and Russell (1987) and translated into Korean by Yoo and Lee (2006). The instrument comprises 24 items, rated using a four-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). It has six subscales assessing attachment, social integration, the opportunity for nurturance, reassurance of worth, reliable alliance, and guidance. Each subscale comprises four items. The total score on social support was calculated by adding the scores of all items and ranged from 24 to 96. Higher scores indicated higher levels of perceived social support. Cronbach's alpha coefficients for the Social support were 0.92 in a prior study (Cutrona & Russell, 1987), 0.94 among Korean male adults (Je, 2014).
post-traumatic stress | one month after the intervention
  PTS was measured using the PCL-5, which was developed by Weathers et al. (2013), revised by Weathers et al. (1993) as per the revised PTSD definition in the DSM-5, and translated into Korean by Kim et al. (2017). The Korean version of the PCL for the DSM-5 (PCL-5-K) contained 20 items, and each scored from 0 (not at all) to 4 (extremely). The score depended on the severity of the symptom caused by stress related to traumatic events during the past month. Possible scores ranged from 0 to 80, with a score of 37 or above indicating a PTSD diagnosis, and higher scores suggesting severe PTSD symptoms (2013). Cronbach's alpha coefficient for the PCL-5-K was .97 among Korean veterans of the Vietnam War (2017).
depression | one month after the intervention
  Depression was assessed using the Center for Epidemiologic Studies Depression Scale (CES-D), developed by Radloff (1997) and translated into Korean by Chon and Rhee (1992). The Korean version of the CES-D contained 20 items rated on a 4-point Likert scale (0 = rarely or never; 3 = all the time), according to how respondents felt during the past week. Possible scores ranged from 0 to 60, with a score of 16 or above indicating depressive symptoms, and higher scores indicating higher levels of depression (1977). Cronbach's alpha coefficient for the Korean CES-D was .89 among Korean adults (1992).
anxiety | one month after the intervention
  Anxiety was measured using the Korean version of the State-Trait Anxiety Inventory (STAI; J. T. Kim & Shin, 1978), originally developed by Spielberger et al. (1970). The STAI comprises 20 items measuring state anxiety, indicating the current degree of anxiety. It has 20 items assessing trait anxiety, indicating the degree of generally feeling anxious. The responses are rated on a four-point Likert scale ranging from 1 (almost never) to 4 (almost always), with the possible range of scores for each type of anxiety being 20-80. Higher scores indicate greater state and trait anxiety. Cronbach's alpha coefficients were 0.87 for state anxiety and 0.86 for trait anxiety in a prior study (S. S. Kim, 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Nursing, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park J, Kim G, Kim S. Exploring trauma recovery in nurses: a text mining and thematic analysis based on Swanson's theory of caring. BMC Nurs. 2025 Mar 12;24(1):279. doi: 10.1186/s12912-025-02757-y. PMID 40075439